CLINICAL TRIAL: NCT00846898
Title: The Effect of Dietary Supplementation of Cinnamon (Cinnamon Cassia) on HbA1c, Blood Pressure and Serum Lipid Measurements in Patients With Type 2 Diabetes Mellitus: a Randomised Placebo Controlled, Double Blind Clinical Trial
Brief Title: Is There a Metabolic Effect of Cinnamon on HbA1c, Blood Pressure and Serum Lipids in Type 2 Diabetes Mellitus?
Acronym: cinnamon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thames Valley University (Other)
Collaborators: Wembley Health Care centre, NHS, UK. (Unknown); Monks Park Primary care centre, NHS UK. (Unknown); Willesden Health centre, NHS, UK. (Unknown)
Responsible Party: Nicky Robinson, Thames Valley University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07/H0717/47
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2011-11-14 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: blood sugar; cholesterol; cinnamon; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cinnamon (Experimental): Subjects in this group will receive cinnamon capsules for 12 weeks period. The 2 g dose of cinnamon will be spread over the day as 500 mg (1 capsule) after breakfast, 1000 mg (2 capsules) after lunch and 500 mg (1 capsule) after dinner. The subjects will be instructed to take the capsules immediately after the meals.
  Interventions: Dietary Supplement: cinnamon 2g per day for 12 weeks
- Control (Placebo Comparator): Subjects in this group will receive placebo capsules (starch flour) for 12 weeks period. The 2 g dose of starch capsules will be spread over the day as 500 mg (1 capsule) after breakfast, 1000 mg (2 capsules) after lunch and 500 mg (1 capsule) after dinner. The subjects will be instructed to take the capsules immediately after the meals.
  Interventions: Dietary Supplement: cinnamon 2g per day for 12 weeks

INTERVENTIONS:
Dietary Supplement: cinnamon 2g per day for 12 weeks — Subjects in intervention group will receive cinnamon capsules for 12 weeks period. The 2 g dose of cinnamon will be spread over the day as 500 mg (1 capsule) after breakfast, 1000 mg (2 capsules) after lunch and 500 mg (1 capsule) after dinner. The subjects will be instructed to take the capsules immediately after the meals.
  Other Names: cinnamon

SUMMARY:
The aim of the study is to assess whether dietary supplementation of cinnamon (cinnamon cassia) has the potential to improve HbA1c, blood pressure and serum lipid measurements in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The study will be conducted for 3 months (12 weeks) with 58 individuals diagnosed with type 2 diabetes mellitus. The randomisation will be carried out by using a randomisation list. Cinnamon bark (cinnamon cassia) and starch flour (placebo) capsules will be purchased from a local pharmaceutical company in UK; these are freely available for over the counter use. Each capsule contained either 500 mg of cinnamon powder or starch flour. The cinnamon and placebo (starch flour) capsules will be packaged in a non transparent plastic bags.

The patients will be randomly allocated into the two groups of:

Group 1: placebo control group Group 2: cinnamon group

Patients in both placebo and cinnamon groups will receive treatment similar to the treatment they would normally receive from their respective NHS or primary care trust for 12 weeks.

Data collection:

After the randomisation the subjects will be scheduled to visit the clinic at 0 weeks, 6 - 7 weeks and 12 weeks from the beginning of the study. During every visit (week 0, weeks 6 - 7 and week 12) a 3-day diet diary will be collected and the intake of total calories, fats, carbohydrates, proteins and fibre will be determined. Compliance with the diet will be monitored by individual discussions at each clinical visit with dietician and compared with the diet diary. The anthropometric measurements of body weight, height, waist and hip circumferences will be measured before the trial (week 0), during the trial (weeks 6 - 7) and after the trial (week 12) period. The recorded clinical measurements of blood profiles include HbA1c level, fasting plasma glucose concentration and serum lipid profiles including serum total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL) and serum triglycerides, systolic and diastolic blood pressures will be measured at the baseline (week 0) and at 12 weeks during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with type 2 diabetes mellitus
2. Aged over 18 years, either sex
3. HbA1c level more than 7%
4. Patients treated only with oral anti-diabetic drugs or diet

Exclusion Criteria:

1. Patients with severe health problems including renal disease, liver disease, cardiovascular disease and other chronic ill health conditions
2. Patients with mental health problems
3. Patients treated with insulin therapy
4. Patients refused to give informed consent
5. Pregnant and lactating women
6. Patients taking cinnamon supplements and other herbal supplements known to be effective

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months

SECONDARY OUTCOMES:
Plasma glucose concentration Plasma lipid profiles (HDL, LDL, Triglycerides and total cholesterol) systolic and diastolic blood pressures. Body Mass Index. Waist circumference. Total calorie intake. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Amalia Tsiami, PhD,MSc,BSc, Study Director — Thames Valley University
Locations (1):
- Brent teaching Primary Care trust (NHS), Wembley, London, United Kingdom